CLINICAL TRIAL: NCT02831543
Title: Clinical Trial to Assess the Efficacy and Safety of Combination Therapy of Motireb 5/100 mg in Functional Dyspepsia Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-REMO-301
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Motireb 5/100 mg t.i.d (Experimental): Motireb 5/100 mg t.i.d + Placebo of Mosapride citrate t.i.d
  Interventions: Drug: Motireb 5/100 mg
- Mosapride citrate t.i.d (Active Comparator): Placebo of Motireb 5/100 mg t.i.d + Mosapride citrate t.i.d
  Interventions: Drug: Mosapride citrate
- Placebo t.i.d (Placebo Comparator): Placebo of Motireb 5/100 mg t.i.d + Placebo of Mosapride citrate t.i.d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Motireb 5/100 mg
  Arms: Motireb 5/100 mg t.i.d
Drug: Mosapride citrate
  Arms: Mosapride citrate t.i.d
Drug: Placebo
  Arms: Placebo t.i.d

SUMMARY:
A phase Ⅲ, multi-center, randomized, double-blinded, placebo and active comparator clinical trial to assess the efficacy and safety of combination therapy of Motireb 5/100 mg in functional dyspepsia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 19 years or older
2. Patient with functional dyspepsia met the ROME III criteria or symptom assessment form

Exclusion Criteria:

1. Patient with peptic ulcer or gastroesophageal reflux disease
2. Patients with previous gastrointestinal surgery
3. Patients with history of gastrointestinal bleeding, mechanical obstruction, perforation
4. Patients with history of gastrointestinal cancer
5. Patients with pancreatic disease (pancreatitis, pancreatic cancer, etc), biliary disease, inflammatory bowel disease, acute gastritis.
6. Patients with Zollinger-Ellison syndrome
7. Patients with irritable bowel syndrome
8. Pregnant or lactating women
9. Patients with hepatic abnormality
10. Patients with renal dysfunction or chronic kidney disease
11. Patients who are judged by the investigators to be unsuitable to participate in the clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The responder ratio of GOS(Global Overall Symptom) | at the 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Kyung-gi, South Korea